CLINICAL TRIAL: NCT00953576
Title: A Phase I/II Trial of Ketoconazole, Hydrocortisone, Dutasteride and Lapatinib (KHAD-L) in Castration Resistant Prostate Cancer With Pre- and Post-therapy Tumor Biopsies
Brief Title: Ketoconazole, Hydrocortisone, Dutasteride and Lapatinib (KHAD-L) in Prostate Cancer
Acronym: KHLAD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study terminated early due to concerns about drug toxicity.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Prostate Cancer Foundation Clinical Research Consortium (Network); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Glenn Bubley, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-374
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
Keywords: castration resistant prostate cancer; KHAD
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ketoconazole; Hydrocortisone; Dutasteride; Lapatinib

STUDY DESIGN:
Intervention Model Description: The Phase I dose escalation schedule was to evaluate up to 4 dose levels of lapatinib as well as one step down dose for ketoconazole (-1). This is not a 'parallel assignment' since this dose escalation design proceeds in sequence not in parallel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I Dose Level 1 (DL1): KHAD+L (250 mg) (Experimental): For the initial four weeks (1 cycle=28 days), participants receive KHAD treatment.
  Ketoconazole: 400 mg orally 3x day Hydrocortisone: 30 mg (a.m.) and 10 mg (p.m.) orally 2x day Dutasteride: 0.5 mg orally 1x day
  Participants start KHLAD on day 29 or d1 of cycle 2/ week 5. Lapatinib: 250 mg orally 1x day
  Participants are treated until unacceptable toxicity, disease progression or withdrawal.
  Interventions: Drug: ketoconazole; Drug: hydrocortisone; Drug: dutasteride; Drug: lapatinib
- Phase I Dose Level 2 (DL2): KHAD+L (500 mg) (Experimental): For the initial four weeks (1 cycle=28 days), participants will receive KHAD treatment.
  Ketoconazole: 400 mg orally 3x day Hydrocortisone: 30 mg (a.m.) and 10 mg (p.m.) orally 2x day Dutasteride: 0.5 mg orally 1x day
  Participants will start KHLAD on day 29 or d1 of cycle 2/ week 5. Lapatinib: 500 mg orally 1x day
  Interventions: Drug: ketoconazole; Drug: hydrocortisone; Drug: dutasteride; Drug: lapatinib
- All Phase I Participants (Experimental): For the initial four weeks (1 cycle=28 days), participants receive KHAD treatment.
  Ketoconazole: 400 mg orally 3x day Hydrocortisone: 30 mg (a.m.) and 10 mg (p.m.) orally 2x day Dutasteride: 0.5 mg orally 1x day
  Participants start KHLAD on day 29 or d1 of cycle 2/ week 5. Lapatinib: according to the established dose escalation schedule
  Participants are treated until unacceptable toxicity, disease progression or withdrawal.
  Interventions: Drug: ketoconazole; Drug: hydrocortisone; Drug: dutasteride; Drug: lapatinib

INTERVENTIONS:
Drug: ketoconazole
  Other Names: Nizoral
Drug: hydrocortisone
  Other Names: Cortef; Hydrocortone
Drug: dutasteride
  Other Names: Avodart
Drug: lapatinib
  Other Names: lapatinib ditosylate; Tyverb

SUMMARY:
The purpose of this research study is to determine the safety of giving ketoconazole, hydrocortisone and dutasteride (KHAD) with lapatinib. Safety is primarily based on dose limiting toxicity (DLT) evaluation at various dose levels (DL). The investigators believe that there is evidence in castrate resistant prostate cancer (CRPC) that two growth factor receptors (EGFR and Her 2/Neu) are increased in prostate cancer (PCa) cells. Both these receptors are turned off by the drug lapatinib. By adding lapatinib, the investigators hope that signaling from the receptors will be turned off and therefore make the participant's cancer more responsive to KHAD treatment.

DETAILED DESCRIPTION:
The current study builds on investigators' KHAD experience by further targeting pathways that may still be enhancing AR activity despite reduced testosterone and DHT. Importantly, studies from several groups have shown that EGFR and Her2/Neu activation can enhance AR signaling and increase AR transcriptional activity in response to low levels of androgens. Evaluation in the clinic and lab has shown that there is increased expression of EGFR or Her2/Neu in CRPC. In addition to upregulation in EGFR and Her2/Neu protein expression, signaling through these receptors may be enhanced in some tumors by increases in growth factor levels or other mechanisms. Based on these results, the investigators suggest that EGFR and Her2/Neu contribute to enhancing AR transcriptional activity especially at low androgen levels. If this hypothesis is correct, then dual blockade of EGFR and Her2/Neu in CRPC should enhance the ability of KHAD to abrogate AR activity. Moreover, as androgens can protect PCa cells from cell death in response to EGFR/Her2/Neu/PI3 kinase pathway inhibition, we propose that KHAD plus lapatinib may be a particularly active combination therapy for CRPC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CRPC with metastatic bone disease. At least one site of metastatic disease must be amenable to a needle biopsy. Bone sites include lumbar vertebrae, pelvic bones and long bones. Excluded sites are thoracic, cervical vertebrae, skull and rib lesions
* Patients may have had a number of previous hormonal therapies including ketoconazole and abiraterone, provided these were discontinued >3 months before starting the trial
* Patients may have had any number of previous cytotoxic therapies
* Castrate resistant disease as defined by PSA working group. Patients must have a rise in PSA on two successive determinations at least one week apart and PSA levels 5ng/ml or greater and testosterone levels <50
* Adequate renal, hepatic and bone marrow function as outlined in protocol
* PTT< 60, INR <1.5NL unless on warfarin therapy
* > 6 month life expectancy
* At least a 4 week interval from previous treatment other than LHRH analog and bisphosphonates. Patients on bicalutamide must have discontinued this medication for at least 6 weeks to be eligible
* Patients receiving bisphosphonate can be maintained on this therapy
* No major surgery or radiation therapy within 4 weeks
* No strontium-89 or samarium-153 therapy within 4 weeks
* ECG showing normal QT interval
* No thromboembolism in past 6 months
* Age > 18 years
* Investigator must check current patient medications against the list of CYP3A4 inhibitors and inducers prior to registration
* Echocardiogram or MUGA demonstrating ejection fraction within institutional normal limits

Exclusion Criteria:

* No previous therapy with lapatinib
* No previous therapy with ketoconazole within 3 months of starting trial
* The use of complementary therapy directed at prostate cancer treatment excluding the following: green tea, commercial multivitamin preparations. Vitamin B complex, C, D, E and multivitamins are permitted if these are being taken at less than 3 times the RDA
* The concomitant use of drugs known to be narrow therapeutic index CYP3A4 substrates are excluded
* Drugs that are sensitive to CYP3A4 substrates are excluded
* Patients taking drugs that may further prolong QT intervals and present a known risk for Torsades de Pointes are excluded.
* Patients who have alcohol or drug dependence currently or in the last 6 months are excluded from this study
* Any other events, other than those defined above, in the opinion of the investigator, may make the patient ineligible for this trial
* No contraindication to biopsy such as bleeding disorders. Patients on anticoagulants such as warfarin must be able to safely stop the drug for a three-day period. Patients may not go on heparin during this time
* No active malignancy other than skin cancer or superficial bladder cancer
* Cardiac disease: congestive heart failure > class II NYHA. Patients must no have unstable angina or new onset angina or myocardial infarction within the past 6 months. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy. Patients must have an ejection fraction within normal limits at the enrolling institution based on an echocardiogram
* Uncontrolled hypertension defined as sustained BP > 160 and diastolic > 100 despite optimal medical management
* Known HIV or chronic Hep B or C
* Thrombolic or embolic events such as CVA within the last 6 months
* Pulmonary hemorrhage or any bleeding event CTCAE Grade 2 or greater within 6 months of first dose of study drug of KHAD
* Serious non-healing wound, ulcer, or bone fracture
* Evidence of history of bleeding diathesis or coagulopathy
* Major surgery or significant traumatic injury within 4 weeks of first study drug of KHAD

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-09-29 (Actual); Primary Completion 2013-04-11 (Actual); Study Completion 2013-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Bubley, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from September 2009 until December 2011.
Groups:
- Phase I Dose Level 1: KHAD+L (250 mg): For the initial four weeks (1 cycle=28 days), participants receive KHAD treatment.
  Ketoconazole: 400 mg orally 3x day Hydrocortisone: 30 mg (a.m.) and 10 mg (p.m.) orally 2x day Dutasteride: 0.5 mg orally 1x day
  Participants start KHLAD on day 29 or d1 of cycle 2/ week 5. Lapatinib: 250 mg orally 1x day
  Participants are treated until unacceptable toxicity, disease progression or withdrawal.
- Phase I Dose Level 2: KHAD+L (500 mg): For the initial four weeks (1 cycle=28 days), participants will receive KHAD treatment.
  Ketoconazole: 400 mg orally 3x day Hydrocortisone: 30 mg (a.m.) and 10 mg (p.m.) orally 2x day Dutasteride: 0.5 mg orally 1x day
  Participants will start KHLAD on day 29 or d1 of cycle 2/ week 5. Lapatinib: 500 mg orally 1x day
  Participants are treated until unacceptable toxicity, disease progression or withdrawal.
Period: Overall Study
Arm/Group | Phase I Dose Level 1: KHAD+L (250 mg) | Phase I Dose Level 2: KHAD+L (500 mg)
Started | 6 | 5
DLT Evaluable (Participants were DLT evaluable if they received 1 cycle of KHLAD and full dose ketoconazole (KHAD).) | 3 | 5
Treated | 4 | 5
Pharmacokinetic (PK) Evaluable (Participants with pre- and post KHLAD day 28 samples.) | 4 | 3
Completed | 4 (One participant enrolled on dose level 1 did not receive full dose ketoconazole and was replaced.) | 4
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Ineligible after Consent | 2 | 0

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 1: KHAD+L (250 mg) | Phase I Dose Level 2: KHAD+L (500 mg) | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Full Range); unit: years] | 66 [51 to 87] | 67 [65 to 69] | 67 [51 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Lapatinib Maximum Tolerated Dose (MTD) [Phase I]
Description: The MTD of lapatinib in combination with KHAD is determined by the number of participants who experience a dose limiting toxicity (DLT) at the various dose levels of lapatinib under evaluation. See subsequent primary outcome measure for the DLT definition. The MTD is defined as the lapatinib dose at which fewer than one-third of patients experience a DLT. If no DLTs are observed, the MTD is not reached and the Recommended Phase II Dose (RP2D) will be based on safety and pharmacokinetic results.
Time Frame: The evaluation for MTD occurred continuously through one cycle of KHLAD treatment (28 days).
Population: The analysis dataset is comprised of all DLT evaluable participants.
Measure: Number; unit: mg 1x daily
Groups:
- All Phase I Participants KHAD+L: For the initial four weeks (1 cycle=28 days), participants receive KHAD treatment.
  Ketoconazole: 400 mg orally 3x day Hydrocortisone: 30 mg (a.m.) and 10 mg (p.m.) orally 2x day Dutasteride: 0.5 mg orally 1x day
  Participants start KHLAD on day 29 or d1 of cycle 2/ week 5. Lapatinib: orally 1x day according to the established dose escalation schedule
  Participants are treated until unacceptable toxicity, disease progression or withdrawal.
Arm/Group | All Phase I Participants KHAD+L
Number analyzed (Participants) | 8
mg 1x daily | NA — While 2 DLTs occurred at DL2, the MTD was not established as DL1 because based on PK analysis, the observed level of lapatinib was well above therapeutic levels which raised sufficient concern to terminate the study.

2. Primary Outcome: Lapatinib Dose Limiting Toxicity (DLT) [Phase I]
Description: A DLT is defined as an adverse event (AE) occurring during the first cycle of KHLAD treatment that are determined to related to the Lapatinib or the combination as follows:
  1. Any Grade 3 or greater non-hematological treatment related (possible, probable, or definite attribution) including diarrhea
  2. Grade 4 or greater for hematological toxicities, regardless of attribution.
  3. Grade 3 skin reactions, pulmonary reactions, regardless of attribution.
Time Frame: The evaluation for DLT occurred continuously through one cycle of treatment (28 days).
Population: The analysis dataset is comprised of all DLT evaluable participants.
Measure: Number; unit: participants with DLT
Arm/Group | Phase I Dose Level 1: KHAD+L (250 mg) | Phase I Dose Level 2: KHAD+L (500 mg)
Number analyzed (Participants) | 3 | 5
participants with DLT | 0 | 2

3. Primary Outcome: Plasma Lapatinib Levels [Phase I]
Description: Plasma lapatinib levels were measured after day 28 of KHLAD treatment. Participants were instructed to fast prior to samples being taken.
Time Frame: After first 28 days of KHLAD treatment
Population: The analysis dataset is comprised of participants who received KHLAD and had an evaluable plasma sample after the first cycle (day 28).
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Phase I Dose Level 1: KHAD+L (250 mg) | Phase I Dose Level 2: KHAD+L (500 mg)
Number analyzed (Participants) | 4 | 3
ng/mL | 731 [416 to 1424] | 1506 [680 to 2186]

4. Secondary Outcome: Grade 3-4 Treatment-Related Adverse Events Rate
Description: All grade 3-4 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 as reported on case report forms were counted to calculate the proportion of participants experiencing at least one treatment-related grade 3 or 4 AE of any type on treatment.
Time Frame: Assessed each cycle throughout treatment. Treatment duration in months was a median (range) of 5.4 months (range 1 day-8.3 months). Thus, AEs were evaluated up to 8.3 months.
Population: The analysis dataset is comprised of all participants who ever started treatment.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Groups:
- Phase I Dose Level 1: KHAD+L (250 mg): For the initial four weeks (1 cycle=28 days), participants receive KHAD treatment.
  For the initial four weeks (1 cycle=28 days), participants will receive KHAD treatment.
  Ketoconazole: 400 mg orally 3x day Hydrocortisone: 30 mg (a.m.) and 10 mg (p.m.) orally 2x day Dutasteride: 0.5 mg orally 1x day Participants will start KHLAD on day 29 or d1 of cycle 2/ week 5. Lapatinib: 250 mg orally 1x day
  Participants are treated until unacceptable toxicity, disease progression or withdrawal.
- Phase I Dose Level 2: KHAD+L (500 mg): For the initial four weeks (1 cycle=28 days), participants will receive KHAD treatment.
  Ketoconazole: 400 mg orally 3x day Hydrocortisone: 30 mg (a.m.) and 10 mg (p.m.) orally 2x day Dutasteride: 0.5 mg orally 1x day
  Participants will start KHLAD on day 29 or d1 of cycle 2/ week 5. Lapatinib: 500 mg orally 1x day
Arm/Group | Phase I Dose Level 1: KHAD+L (250 mg) | Phase I Dose Level 2: KHAD+L (500 mg)
Number analyzed (Participants) | 4 | 5
proportion of participants | 0 [0.0 to 0.451] | 0.40 [0.076 to 0.811]

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment. Median (range) treatment duration (months) for dose level 1: 5.5 (1.8-8.3) and dose level 2: 5.4 (0.2-17.9). Thus, AEs were followed up to 17.9 months.
Description: The analysis dataset is comprised of all participants who ever started treatment. Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment attribution of possibly, probably or definitely and grade 3 or higher. All remaining events regardless of treatment attribution were classified as Other AEs. No further data is available to specify classification of other beyond the general term.
Arm/Group | Phase I Dose Level 1: KHAD+L (250 mg) | Phase I Dose Level 2: KHAD+L (500 mg)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/5
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 1: KHAD+L (250 mg) (N=4) | Phase I Dose Level 2: KHAD+L (500 mg) (N=5)
Cardiac-other (Cardiac disorders) | 0 | 1 — AE connected with grade 3 or higher EKG changes
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 1: KHAD+L (250 mg) (N=4) | Phase I Dose Level 2: KHAD+L (500 mg) (N=5)
ALT, SGPT (Investigations) | 0 | 1
Amylase (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
AST, SGOT (Investigations) | 1 | 2
Back, pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Cardiac-other (Cardiac disorders) | 2 | 2
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Creatinine (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Edema limb (General disorders) | 0 | 2
Endocrine-other (Endocrine disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Fatigue (General disorders) | 3 | 5
Fever w/o neutropenia (General disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
GI-other (Gastrointestinal disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Hot flashes (Vascular disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
Incontinence, anal (Gastrointestinal disorders) | 0 | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1 | 0
Infection w/ gr3-4 neut, urinary tract (Infections and infestations) | 0 | 1
Infection w/ unk ANC ungual (nails) (Infections and infestations) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Lip, pain (Gastrointestinal disorders) | 1 | 0
Lipase (Investigations) | 1 | 0
Lymphatics-other (Blood and lymphatic system disorders) | 0 | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 0
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Neuropathy-motor (Nervous system disorders) | 1 | 0
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 0 | 1
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain-other (General disorders) | 0 | 2
QTc interval (Investigations) | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Rectum, hemorrhage (Gastrointestinal disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal/GU-other (Renal and urinary disorders) | 1 | 1
Rigors/chills (General disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Skin-other (Skin and subcutaneous tissue disorders) | 2 | 1
Stoma, GI hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Testicle, pain (Reproductive system and breast disorders) | 0 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1 | 0
Urine color (Renal and urinary disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Weight gain (Investigations) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early due to concern of exposure levels observed in PK analyses for the drug under investigation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No